CLINICAL TRIAL: NCT06304246
Title: Is Preoperative Serum Asprosin Level Associated With Preoperative Pain Threshold and Postoperative Analgesic Consumption in Patients Undergoing Cesarean Section Surgery?"
Brief Title: The Relationship Between Preoperative Serum Asprosin Level and Postoperative Analgesic Consumption in Patients Undergoing Caesarean Section
Status: Not yet recruiting | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Sibel Ozcan, Associate Professor, Firat University
Other Study IDs: FU-S.OZCAN 001
Record Dates: First submitted 2024-02-26; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Obstetric Pain; Cesarean Section; Postoperative Pain
Keywords: postoperative pain; cesarean section; pain threshold; obstetric pain
MeSH Terms: conditions — Labor Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Labor Pain Group (LPG): LPG; pregnant women who will undergo emergency C-section with labor pain. Labor pain will be defined as having 3 or more regular uterine contractions in 20 minutes or >120 Montevideo units of uterine performance observed during non-stress testing (NST) conducted at the Obstetrics Clinic.
  Interventions: Other: Measurement Pain Threshold; Other: Measurement of Serum Asprosin
- No Pain Group (NPG): NPG; pregnant women who will undergo elective C-section without labor pain.
  Interventions: Other: Measurement Pain Threshold; Other: Measurement of Serum Asprosin

INTERVENTIONS:
Other: Measurement Pain Threshold — Measurement Pain Threshold: Manual dolorimetry will be used to assess the pain threshold in the non-dominant hand of patients in the preoperative waiting room prior to spinal anesthesia. The dolorimeter head will be placed vertically on the wrist of the non-dominant hand, and pressure will be applied with increments of 1 kg/cm2/s. The pressure applied when the patient perceives pain will be recorded in kg/cm2. The measurement will be repeated three times for each patient, and the average will be recorded as the pain threshold value.
Other: Measurement of Serum Asprosin — Measurement of Serum Asprosin: For serum asprosin measurements, blood will be drawn in the preoperative waiting room before the application of spinal anesthesia. The blood samples will be centrifuged, and the serum will be stored at -20°C to measure serum asprosin levels. After all patient blood is collected, serum asprosin will be evaluated with a commercially available double antibody sandwich enzyme-linked immunosorbent assay (ELISA) kit.

SUMMARY:
Adipokines are bioactive substances secreted from adipose tissue and have various functions on appetite, energy, lipid, carbohydrate metabolism, regulation of blood pressure, and inflammation. One of these is asprosin, discovered in 2016, which is secreted from white adipose tissue. It has been shown that the level of asprosin encoded by the Fibrillin 1 gene can vary in metabolic syndrome associated with obesity, diabetes, and insulin resistance . Some adipokines such as leptin, adiponectin, or resistin are found in increasing levels in the blood and placenta as pregnancy progresses. The detection of high concentrations of adipokines in cord blood has shown that they play an important role in fetal development and metabolism, can interfere with placental development, and affect pregnancy outcomes and fetal growth. Adipokines associated with appetite, energy, lipid, and carbohydrate metabolism have been shown to be effective in modulating pain in recent years. High levels of leptin have been shown to be associated with decreased preoperative pain threshold and increased postoperative analgesic consumption. Recent studies have indicated that asprosin also exhibits analgesic effects in neuropathic pain models and may have clinical benefits in alleviating chronic pain associated with diseases and injuries originating from peripheral structures.

It is known that one of the most important factors affecting mothers' approach to anesthesia technique in Cesarean section is their fear of intraoperative and postoperative pain. Almost one in five patients experiences severe acute pain after Cesarean section. Pain can be perceived differently by patients, and even with the same anesthesia technique, some patients may experience more severe pain. Patients' perception of pain is influenced by many factors such as pain threshold, mood, hormonal balance, central sensitization, and genetic factors.

We hypothesized that the increased preoperative serum asprosin levels might be associated with increased acute labor pain and that asprosin levels might lead to increased analgesic use in the postoperative period. Additionally, we assumed that patients could alter their preoperative pain threshold and report higher pain scores after surgery due to hyperalgesia caused by high asprosin levels.

In this study, we aimed to investigate preoperative serum asprosin levels in patients undergoing Cesarean section with and without acute labor pain and to determine whether there is a relationship between preoperative asprosin levels and postoperative analgesic use.

DETAILED DESCRIPTION:
Subjects: A total of 50 pregnant women, who are scheduled for elective cesarean section and request spinal anesthesia for cesarean surgery, will be enrolled in the study. Patients will be divided into two groups as follows: the labor pain group (LPG, pregnant women who will undergo emergency C-section with labor pain) and the no pain group (NPG, pregnant women who will undergo elective C-section without labor pain). Labor pain will be defined as having 3 or more regular uterine contractions in 20 minutes or >120 Montevideo units of uterine performance observed during non-stress testing (NST) conducted at the Obstetrics Clinic.

Patients under the age of 18, those with preeclampsia, eclampsia, gestational diabetes, or hypertension, patients with abnormal pregnancies, systemic diseases, or diabetes will be excluded from the study.

Patient characteristics such as age, height, weight, body mass index, ASA and Mallampati scores, gestational week, previous cesarean section count, existing medical conditions, family history, smoking and alcohol use status, and pregnancy-related conditions and complications will be recorded.

Measurement of Serum Asprosin: For serum asprosin measurements, blood will be drawn in the preoperative waiting room before the application of spinal anesthesia. The blood samples will be centrifuged, and the serum will be stored at -20°C to measure serum asprosin levels.

Measurement Pain Threshold: Manual dolorimetry will be used to assess the pain threshold in the non-dominant hand of patients in the preoperative waiting room prior to spinal anesthesia. The dolorimeter head will be placed vertically on the wrist of the non-dominant hand, and pressure will be applied with increments of 1 kg/cm2/s. The pressure applied when the patient perceives pain will be recorded in kg/cm2. The measurement will be repeated three times for each patient, and the average will be recorded as the pain threshold value.

Postoperative Pain Severity: Postoperative pain severity will be evaluated using the visual analog scale (VAS). Before the evaluation, patients will be informed about the VAS and its pain scoring system, which ranges from 0 (no pain) to 10 (extreme pain). All patients will be monitored carefully, and their VAS scores will be recorded at 1, 2, 4, 6, 12, and 24 h postoperatively.

Consumption of Postoperative Analgesic: For postoperative analgesia, patients will be provided with tramadol-based patient-controlled analgesia. The time of the first analgesic requirement and the total amount of analgesic used after 24 hours will be recorded.

Statistics: Continuous variables will be expressed as mean ± standard deviation. The normal distribution of numerical variables will be checked using the Kolmogorov-Smirnov test. Independent sample t-test will be used for comparing two independent groups when data are normally distributed, and the Mann-Whitney U test will be used when data are not normally distributed. Spearman's rho correlation coefficient will be used to examine the relationships between asprosin levels, pain threshold, VAS score, and analgesic consumption. Multiple regression analysis will be performed to examine the effects of asprosin levels and group variables on analgesic consumption and pain threshold. P <0.05 will be considered statistically significant for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women who are scheduled for elective cesarean section and request spinal anesthesia for cesarean surgery,

Exclusion Criteria:

* Being under the age of 18
* Having an abnormal pregnancy with preeclampsia, eclampsia, gestational diabetes, or hypertension
* Having a comorbid desease, systemic diseases, cardiovascular disease
* Having diabetes, obesity, or infection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: Pregnant women who applied to the Obstetrics and Gynecology Clinic at Fırat University Hospital and were planned for elective cesarean section and requested spinal anesthesia for cesarean section will participate.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Preoperative Asprosin Level | Before the application of spinal anesthesia
  Serum asprosin measurements, blood will be drawn in the preoperative waiting room before the application of spinal anesthesia.
Postoperative Pain | postoperative 1st hour, 2nd hour, 4th hour, 6th hour, 12th hour and 24th hour
  Postoperative pain will be assessed using visual analogous scale (VAS) ranging from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Postoperative analgesic consumption | First 24 hours postoperatively
  Patients will be provided with tramadol-based patient-controlled analgesia. The time of the first analgesic requirement and the total amount of analgesic used after 24 hours will be recorded.

IPD SHARING:
Plan to Share IPD: Undecided
I will decide after the study is completed.